CLINICAL TRIAL: NCT07111988
Title: Valbenazine in Obsessive-compulsive Disorder: A Randomized Double-blind Placebo-controlled Crossover Trial
Brief Title: Valbenazine in Obsessive Compulsive Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB25-0568
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — valbenazine

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled crossover trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valbenazine followed by placebo (Other): Following baseline measures, 50% of subjects will receive valbenazine (initially 40mg per day for 2 weeks and then 80mg per day for 4 weeks). This will be followed by a 2-week washout period and then 6 weeks of being assigned to the other agent. Participants will be assessed at baseline and every 2 weeks during the remainder of the study period.
  Interventions: Drug: Valbenazine
- Placebo followed by valbenazine (Other): Following baseline measures, 50% of subjects will receive inactive placebo for 6 weeks. This will be followed by a 2-week washout period and then 6 weeks of being assigned to the other agent (initially 40mg per day for 2 weeks and then 80mg per day for 4 weeks). Participants will be assessed at baseline and every 2 weeks during the remainder of the study period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valbenazine — Selective vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: Ingrezza
  Arms: Valbenazine followed by placebo
Drug: Placebo — Pill that contains no medicine
  Other Names: No other names
  Arms: Placebo followed by valbenazine

SUMMARY:
The primary aim of the study is to examine the efficacy and safety of valbenazine in adults with moderate to severe obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
The primary aim of the study is to examine the efficacy and safety of valbenazine in adults with moderate to severe obsessive-compulsive disorder (OCD). Subjects will either receive double-blind valbenazine or inactive placebo for 6 weeks. This will be followed by a 2-week washout period and then 6 weeks of being assigned to the other agent (valbenazine or placebo). The hypothesis to be tested is that valbenazine will significantly improve symptoms of OCD compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65 years
2. Primary diagnosis of obsessive compulsive disorder (OCD)
3. Yale Brown Obsessive Compulsive Scale (Y-BOCS) score of at least 21 at baseline (moderate or higher severity)
4. Ability to understand and sign the consent form

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity Rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
4. History of psychosis or bipolar disorder based on DSM-5 criteria
5. Alcohol/substance use disorder and/or illegal substance use based on urine toxicology
6. Initiation of psychological interventions within 3 months of screening (those who are continuing with CBT will be included)
7. Use of any new psychotropic medication within 3 months of study entry (stable doses of psychotropics will be allowed)
8. Major cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent
9. Abnormal liver function tests at baseline (greater than 2x the upper limit of normal)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | Baseline to week 14
  A clinician-administered scale assessing OCD severity that will be used at all 8 visits. Total scores range from 0-50. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB) cognitive testing | Baseline to week 14
  Objective neuropsychological tasks, including the Tower of London Task, the Intra-dimensional/Extra-dimensional Set Shift (IED) task, the Cambridge Gambling Task (CGT), the Spatial Working Memory (SWM) task, and the Rapid Visual Information Processing (RVP) task, that will be administered pre- and post-pharmacological trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No